CLINICAL TRIAL: NCT03149237
Title: Partners-based HIV Treatment for Sero-concordant Couples Attending Antenatal Care
Brief Title: Partners-based HIV Treatment for Couples Attending Antenatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carolyn Audet, Assistant Professor of Health Policy, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 170365; R01MH113478-01 (NIH)
Record Dates: First submitted 2017-05-03; First posted 2017-05-11 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: Mozambique; Couples-based services; HIV/AIDS; Ante-natal Care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The 12 clinics randomly assigned to the intervention arm will receive a combination of community and clinical services, including: (1) ANC-based couples HIV testing, couples-based treatment enrollment, and clinical care for sero-concordant HIV+ expectant couples; (2) couple-centered treatment in the post-partum period; (3) couples-based education and skills building during the ANC and post-partum period; and (4) treatment continuity support by expert-patient (peer) navigators selected among couples who have successfully navigated EMTCT. The 12 clinics randomized to the control arm will continue to provide standard of care EMTCT services that include: standard HoPS male engagement (male invitation to ANC services and couples HIV testing), opt-out rapid HIV testing of all pregnant women attending ANC, HIV-specific counseling and support for all women who test positive, provision of cotrimoxazole prophylaxis, and universal ART, as per option B+ guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The 12 clinics randomized to the control arm will continue to provide standard of care (SOC) EMTCT services that include: standard HoPS male engagement (male invitation to ANC services and couples HIV testing), opt-out rapid HIV testing of all pregnant women attending ANC, HIV-specific counseling and support for all women who test positive, provision of cotrimoxazole prophylaxis, and universal ART, as per option B+ guidelines.
- Couples-based Services (Experimental): The 12 clinics randomly assigned to the intervention arm will receive a combination of community and clinical EMTCT services, including: (1) ANC-based couples HIV testing, couples-based treatment enrollment, and clinical care for sero-concordant HIV+ expectant couples; (2) couple-centered treatment in the post-partum period at the EID clinic; (3) couples-based education and skills building during the ANC and post-partum period; and (4) treatment continuity support by expert-patient (peer) navigators selected among couples who have successfully navigated EMTCT.
  Interventions: Behavioral: Couples-based services

INTERVENTIONS:
Behavioral: Couples-based services — Couples-based services, including treatment, counseling and peer mentoring in the community.
  Arms: Couples-based Services

SUMMARY:
The purpose of this R01 proposal is to evaluate the clinical impact, hypothesized mechanisms of behavior change, and cost-effectiveness of a partners-focused integrated elimination of mother-to-child transmission of HIV (EMTCT) package comprised of: 1) antenatal care-based couples HIV testing, ART enrollment, and care for sero-concordant HIV+ expectant couples; (2) Couples-based treatment in the post-partum period; (3) Couple-based education and skills building; and (4) Treatment continuity with the support of expert-patient (peer) supporters from couples who have successfully navigated EMTCT. This innovative approach to scaling up EMTCT services, if proven feasible and effective, will be adopted in President's Emergency Plan for AIDS Relief (PEPFAR) programs to accelerate progress toward EMTCT and helping families with HIV infection live long, healthy lives.

DETAILED DESCRIPTION:
In severely resource-limited rural settings, scale-up of services to eliminate mother-to-child transmission of HIV (EMTCT) has failed to provide effective HIV testing and antiretroviral therapy (ART) coverage for women in highest prevalence southern African regions. All HIV-infected pregnant women are now eligible for life-long antiretroviral therapy (ART) (Option B+), but retention among women enrolled through Option B+ programs remains sub-optimal. In sub-Saharan Africa (SSA) it is common for women to require male partner approval to access and remain engaged in HIV-related health services. Despite the likelihood that male involvement would improve program coverage and adherence, the evidence base for effective interventions to involve male partners in HIV testing and treatment through antenatal care (ANC) point of care is very limited. Furthermore, whether such strategies are indeed cost-effective for improving outcomes of HIV-diagnosis and treatment in pregnancy is unknown. This proposal seeks to address these key gaps in the evidence base and guide scale-up by evaluating a promising male engagement intervention ("Homens para Saúde" (HoPS)+ [Men for Health]) targeting EMTCT in Mozambique through a clinic-randomized trial. This study will engage 24 ANC clinics; 12 intervention and 12 standard of care, with 45 HIV-infected couples per clinic where currently >60% of couples attend their first ANC visit together. The planned intervention addresses social-structural and cultural factors influencing EMTCT through the creation of couples-centered integrated HIV services, including: (1) ANC-based couples HIV testing, ART enrollment, and care for sero-concordant HIV+ expectant couples; (2) Couple-based treatment in the post-partum period; (3) Couple-based education and skills building; and (4) Treatment continuity with the support of expert-patient (peer) supporters from couples who have successfully navigated EMTCT. Given that 8.0% of all pregnant women and 7.2% of their partners tested HIV-positive during ANC visits in 2015 (FGH monitoring and evaluation [M&E] data), the investigators pioneering work in Mozambique's rural Zambézia province suggests that innovative strategies are essential to engaging HIV-infected male partners in antenatal care (ANC) in order to achieve EMTCT and to improve substantially the health of the mothers. This team of Mozambican and U.S. investigators has a proven record of international HIV research success and they have specific recent experience with EMTCT cluster randomized trials, male-engagement in ANC services, and cost-effectiveness analysis of HIV programs. The specific aims of this study are: (1) To implement and evaluate the impact of male-engaged, couples-centered services on retention in care, adherence to ART, and early infant diagnosis among HIV+ pregnant women and their HIV+ male partners through a cluster-randomized control trial (RCT); (2) To investigate the impact of HoPS+ on hypothesized mechanisms of change; and (3) To use validated simulation models to evaluate cost-effectiveness of the HoPS+ intervention with the use of programmatic provincial monitoring and evaluation data and data from the trial results.

ELIGIBILITY:
Inclusion Criteria:

* Couples, one HIV+ pregnant woman and her infected male partner, will be eligible to participate if the woman's due date is >2 weeks from enrollment. Both persons must also be 18 years or older, able to give consent, willing to consent to an infant record search, and must agree to enroll in ART together.

Exclusion Criteria:

* Couples will not be eligible to participate in the study if the woman is not pregnant, if both persons are not HIV+, if either person is younger than 18 years, if one member of the couple is unwilling to enroll in ART or consent to the infant record search, or if one member of the couple is unable to give consent due to mental limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2160 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Graves, MPH, BSN, Study Director — Vanderilt University
Locations (1):
- Minisitry of Health Health Facility, Pebane, Zambezia Province, Mozambique

IPD SHARING:
Plan to Share IPD: No
After the study is completed and the results published, the investigators will upload de-identified data to ICPSR.

REFERENCES:
- [Derived] Audet CM, Graves E, Shepherd BE, Prigmore HL, Brooks HL, Emilio A, Matino A, Paulo P, Diemer MA, Frisby M, Sack DE, Aboobacar A, Barreto E, Van Rompaey S, De Schacht C. Partner-Based HIV Treatment for Seroconcordant Couples Attending Antenatal and Postnatal Care in Rural Mozambique: A Cluster Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2024 Jul 1;96(3):259-269. doi: 10.1097/QAI.0000000000003440. PMID 38905476
- [Derived] Sack DE, Frisby MB, Diemer MA, De Schacht C, Graves E, Kipp AM, Emilio A, Matino A, Barreto E, Van Rompaey S, Wallston KA, Audet CM. Interpersonal reactivity index adaptation among expectant seroconcordant couples with HIV in Zambezia Province, Mozambique. BMC Psychol. 2020 Aug 28;8(1):90. doi: 10.1186/s40359-020-00442-0. PMID 32859272

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 24 health facilities in Mozambique. It began in November of 2017 and was completed in December 2020
Units Other Than Participants: 24
Period: Overall Study
Arm/Group | Standard of Care | Couples-based Services
Started | 1108; 12 24 | 1052; 12 24
Completed | 1104; 12 24 | 1047; 12 24
Not Completed | 4; 0 24 | 5; 0 24
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Couples-based Services | Total
Number analyzed (Participants) | 1104 | 1047 | 2151
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (5.9) | 26.2 (5.8) | 26.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 552 | 525 | 1077
  Male | 552 | 522 | 1074
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1104 | 1047 | 2151
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mozambique | 1104 | 1047 | 2151
Education [Count of Participants; unit: Participants]
  None | 188 | 120 | 308
  Some/completed primary | 717 | 726 | 1443
  more than primary | 199 | 201 | 400

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Time on Medication Among Pregnant Women
Description: Specifically, every patient is given 30 days to pick up their medication, with a grace period of 5 days. If a patient picks up medication more than 35 days from their last pick-up, then they will be considered not on their medication from day 30 until the day of their next pick-up, at which time they will be assumed to be on medication again; this will be calculated over the course of the one-year follow-up.
Time Frame: 12 months
Population: This is the primary analysis among women
Measure: Mean (Standard Deviation); unit: proportion of days with medicaiton
Arm/Group | Standard of Care | Couples-based Services
Number analyzed (Participants) | 552 | 525
proportion of days with medicaiton | 0.67 (0.26) | 0.66 (0.27)

2. Primary Outcome: Proportion of Days With Medication Among Male Partner
Description: Proportion of days with medication (based on date of pick up and the number of pills provided by the pharmacy) among male partners
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: proportion of days with medicaiton
Arm/Group | Standard of Care | Couples-based Services
Number analyzed (Participants) | 552 | 522
proportion of days with medicaiton | 0.47 (0.31) | 0.55 (0.29)

ADVERSE EVENTS:
Time Frame: During the 18 months the individual was in the study
Arm/Group | Standard of Care | Couples-based Services
All-Cause Mortality (participants affected / at risk) | 25/1104 | 23/1047
Serious Adverse Events (participants affected / at risk) | 0/1104 | 0/1047
Other Adverse Events (participants affected / at risk) | 0/1104 | 0/1047

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT03149237/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT03149237/ICF_000.pdf